CLINICAL TRIAL: NCT02512237
Title: A Phase 1, Multicenter, Open-label, Multiple Dose-escalation Study of ARX788, Intravenously Administered as a Single Agent in Subjects With Advanced Cancers With HER2 Expression
Brief Title: A Dose-escalation Study of ARX788, IV Administered in Subjects With Advanced Cancers With HER2 Expression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replace with a new trial
Sponsor: Zhejiang Medicine Co., Ltd. (Industry)
Collaborators: Ambrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZMC-ARX788-101; Universal Trial Number (UTN) (Registry Identifier: U1111-1173-5221)
Record Dates: First submitted 2015-06-22; First posted 2015-07-30 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasms; Stomach Neoplasms
Keywords: HER2; breast cancer; ADC; antibody drug conjugate; elevated HER2 expression
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1a: Dose-Escalation (Experimental): Six cohorts with escalated dose levels of ARX788 at 0.33 mg/kg, 0.66 mg/kg, 1.3 mg/kg, 2.2 mg/kg, 2.9 mg/kg and 3.8 mg/kg will be administered every 3 weeks via intravenous infusion to determine the MTD.
  Interventions: Drug: ARX788
- Phase 1b: Dose-evaluation 1 (Experimental): Breast cancer subjects with high HER2 expression, categorized as ISH positive or IHC3+, will be administered with ARX788 at MTD every 3 weeks via intravenous infusion.
  Interventions: Drug: ARX788
- Phase 1b: Dose-evaluation 2 (Experimental): Breast cancer subjects with mid/low HER2 expression, categorized as ISH negative AND IHC2+, will be administered with ARX788 at MTD every 3 weeks via intravenous infusion.
  Interventions: Drug: ARX788
- Phase 1b: Dose-evaluation 3 (Experimental): Gastric cancer subjects with high HER2 expression, categorized as ISH positive or IHC3+, will be administered with ARX788 at MTD every 3 weeks via intravenous infusion.
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — ARX788, an antibody drug conjugate

SUMMARY:
This is a 2-part, Phase 1 FIH study with Phase 1a designed to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) in subjects with metastatic cancers with a human epidermal growth factor receptor 2 (HER2) test result that is in situ hybridization (ISH) positive (+) or immunohistochemistry (IHC) 3+ or 2+, and Phase 1b designed to assess anticancer activity and safety in three expansion cohorts: two different advanced breast cancer expansion cohorts (namely, for tumors that test as HER2 ISH positive or IHC3+ and for tumors that test as HER2 ISH negative with IHC 2+), and one advanced gastric cancer expansion cohort (for tumors that test as HER2 ISH positive or IHC3+).

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy >12 weeks.
2. BMI is between 18 to 32 kg/m2
3. Subjects whose advanced cancer has failed treatment or whose cancer has progressed following available standard therapy or for whom such therapy is not acceptable to the subject. Subjects whose tumor tissue local laboratory results are HER2 ISH positive or IHC3+ must have been previously treated with a HER2 targeting therapy (e.g. trastuzumab, in the country or region where such therapies are available and part of standard of care), or have failed SOC therapy. Subjects who have been previously treated with a HER2 targeting therapy such as trastuzumab or ado-trastuzumab emtansine are eligible.
4. Disease measurability: Phase 1a: measureable or non-measureable disease; Phase 1b: disease must be measureable (per RECIST v1.1) (subjects with non-measureable disease are not eligible for Phase 1b).
5. Histopathologic evidence of breast cancer based upon pathologist's report.
6. Tumor tissue local laboratory HER2 testing results (clinical pathology report) based on FDA or other regulatory agency approved, validated or commercially available IHC or ISH HER2 assay. Pre-screening for HER2 is allowed only for subjects with breast and gastric cancer, where applicable. Subjects with other types of cancer must have previously tested for HER2 status by HER2 IHC or ISH assay. 1) Phase 1a: ISH positive or IHC 2+ or 3+. 2) Phase 1b: Cohort 1: advanced breast cancer, ISH positive or IHC 3+; Cohort 2: advanced breast cancer, ISH negative with IHC 2+; and Cohort 3: advanced gastric cancer, ISH positive or IHC 3+.
7. Local pathology laboratory determination of HER2 status will be accepted, provided that the local laboratory is an accredited site for HER2 testing. In Phase 1b, if the local laboratory was not accredited at the time of testing, an adequate tumor tissue sample is required for central pathology laboratory HER2 testing. The tissue sample may be provided as 10 pre-cut unstained slides or a tumor block.
8. Eastern Cooperative Oncology Group Performance Status of 0 to 1.
9. Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade 0 or 1 as per the NCI-CTCAE v 4.03.
10. The last dose of prior anticancer therapy must have been administered at least 28 days prior to the first dose of the IMP.
11. Adequate bone marrow function defined by absolute neutrophil count of ≥1.5×109/L, platelet count of ≥100.0×109/L, and hemoglobin of ≥9.0 g/dL.
12. Adequate hepatic function defined by serum total bilirubin ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase/alanine aminotransferase ≤2.5 × ULN (or ≤5 × ULN in subjects with liver metastases).
13. Adequate renal function assessed by serum creatinine within reference lab normal limits and creatinine clearance (by Chronic Kidney Disease Epidemiology [CKD-EPI] Collaboration equation) ≥60 mL/min.
14. Adequate cardiac function as assessed by cardiac troponin I within normal range; left ventricular ejection fraction ≥ 50% or institutional lower limit of normal; cumulative anthracycline dose <360 mg/m2 doxorubicin or equivalent.
15. Willing and able to understand and sign an informed consent inform and to comply with all aspects of the protocol.
16. Female subjects must be surgically sterile, or have a monogamous partner who is surgically sterile, or at least 2 years postmenopausal, or who commits to use an acceptable form of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 3 months following the last dose of study treatment.
17. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study.

Exclusion Criteria: Any subject who meets any of the following criteria should be excluded from the study:

1. History of allergic reactions to any component of the ARX788.
2. 2. History of seizure disorder.
3. History of unstable central nervous system (CNS) metastases or seizure disorder related to the malignancy; however, those subjects who were treated for prior CNS metastases and who are asymptomatic may participate in the study as long as they are not receiving treatment with steroids.
4. History of congestive heart failure, unstable angina pectoris, unstable atrial fibrillation, or cardiac arrhythmia.
5. Grade 2 to 4 peripheral neuropathy (NCI CTCAE v 4.03).
6. Non-manageable electrolyte imbalances including hypokalemia, hypocalcemia, or hypomagnesemia (Grade 2 or greater based on NCI CTCAE v 4.03).
7. Any uncontrollable intercurrent illness, infection, or other conditions that could limit study compliance or interfere with assessments.
8. Exposure to any other investigational or commercial anticancer agents or therapies administered with the intention to treat malignancy within 28 days before the first dose of the IMP.
9. Significant surgical intervention within 21 days of the first dose of the IMP or with ongoing post-operative complications if more than 21 days.
10. Radiotherapy administrated less than 21 days prior to the first dose of the IMP, or localized palliative radiotherapy administered less than 7 days prior to the first dose of the IMP, or radiotherapy induced toxicity of Grade 2 or greater based on NCI CTCAE v 4.03.
11. Pregnancy or breast feeding.
12. Refusal to use effective methods of contraception (see inclusion criteria for details).
13. Legal incapacity/limited legal capacity for providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ARX788 | 12 months
  Determine highest dose level at which less than 2 of 6 subjects experience a dose limiting toxicity.

SECONDARY OUTCOMES:
Number of subjects with Adverse Events | 30 months
  Safety and tolerability of ARX788 as measured by all adverse events, hematology, blood chemistry, vital signs, electrocardiogram, and physical exam.
Area under the plasma concentration versus time curve (AUC) of ARX788 after infusion | 30 months
  Pharmakokinetic characteristics of ARX788 for infusion Cycle 1 and Cycle 3
Half-life of ARX788 after infusion | 30 months
  Pharmakokinetic characteristics of ARX788 for infusion Cycle 1 and Cycle 3
Number of participants with tumor response to ARX788 administration | 18 months
Number of subjects developed anti-ARX788 antibody | 30 months
  Immunogenicity profile assessment

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Epworth Healthcare, Richmond, Victoria
- New Zealand (3):
  - Auckland City Hospital, Grafton, Auckland
  - Wellington Hospital, Newtown, Wellington Region
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: No